CLINICAL TRIAL: NCT00549159
Title: Multicenter Randomized Clinical Trial to Evaluate the Safety and Effectiveness of Cavaterm TM Thermal Balloon Endometrial Ablation in Women With Dysfunctional Uterine Bleeding Compared to Transcervical Resection of the Endometrium (TCRE)
Brief Title: CavatermTM vs TCRE in Women With DUB
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Pnn Medical A/S (Industry)
Responsible Party: Gediminas Puras, Clinical Trial Manager, Pnn Medical A/S
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2006-0026-06 dd20070920
Record Dates: First submitted 2007-10-24; First posted 2007-10-25 (Estimated); Last update posted 2008-05-22 (Estimated); Status verified 2008-05

CONDITIONS: Dysfunctional Uterine Bleeding
Keywords: menorrhagia; dysfunctional uterine bleeding; endometrial ablation
MeSH Terms: conditions — Metrorrhagia; Menorrhagia

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Cavaterm (Experimental)
  Interventions: Device: Thermal Balloon Endometrial Ablation
- TCRE (Active Comparator): Transcervical resection of the endometrium
  Interventions: Device: Transcervical Resection of the Endometrium

INTERVENTIONS:
Device: Thermal Balloon Endometrial Ablation — Thermal balloon endometrial ablation
  Arms: Cavaterm
Device: Transcervical Resection of the Endometrium — Transcervical resection of the endometrium
  Arms: TCRE

SUMMARY:
The purpose of study is to compare the treatment success in the study groups.

DETAILED DESCRIPTION:
Study success will be defined as reduction of uterine bleeding evaluated by number of patients obtaining amenorrhea, hypomenorrhea or eumenorrhea quantified by PBLAC<75.

ELIGIBILITY:
Inclusion Criteria:

* Willingness and adequate mental capacity to sign written, informed consent
* Willingness to adhere to study plan regarding control visits and recording of PBLAC
* > 30 years old
* Pre-menopausal as determined by FSH ≤30
* Agree not to use hormonal contraception or any other intervention for bleeding during study
* Suitable for local and/or general anesthesia
* A minimum PBLAC score of ≥ 150 for three months prior to study enrollment; OR PBLAC score 150 for one month for women who 1) had at least 3 (documented) prior months of failed medical therapy; 2) had a contraindication to medical therapy; or 3) refused medical therapy
* Uterine cavity sound measurement ≥ 4 cm and ≤ 10 cm.

Exclusion Criteria:

* Presence of bacteriaemia, sepsis, or other active systemic infection
* Active pelvic inflammatory disease
* Clotting defects or bleeding disorders
* Unwillingness to use a non-hormonal birth control post-ablation
* Desire for future fertility
* Abnormal cavity as confirmed by hysteroscopy, transvaginal ultrasound or HSG e.g. large fibroids, septum etc. Small submucosal fibroids defined as < 2 cm are in this context not considered abnormal.
* Any condition leading to possible uterine wall weakness with total wall thickness < 15 mm e.g. at c.section, postmyomectomy scars etc. In case of uniform uterine wall the wall thickness at the fundus should be measured.
* Premalignant or malignant uterine condition within the last five years as confirmed by histology
* Pregnancy
* Cervical length > 6 cm.
* Uterine cavity >30 ml defined as balloon can be filled with 30ml glucose solution without reaching the target pressure of 240 mmHg. (These patients may still be treated as planned but will be withdrawn from the study and their data will be analysed separately. The patients will be recorded as screening failures).
* Previous ablation or subtotal hysterectomy

Ages: 30 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 158 (Estimated)
Dates: Start 2007-10; Primary Completion 2009-10 (Estimated); Study Completion 2009-10 (Estimated)

PRIMARY OUTCOMES:
Reduction of uterine bleeding evaluated by number of patients obtaining amenorrhea, hypomenorrhea or eumenorrhea quantified by PBLAC<75 | 12 months

SECONDARY OUTCOMES:
SF-12, Patients Wishes and Expectations questionnaire, adverse events, need for re-treatment | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Yanhong Yu, Prof., Principal Investigator — Guangzhou Southern Hospital
Locations (2):
- China (2):
  - Zhu Jiang Hospital, Guangzhou, Guangdong
  - Guangzhou Southern Hospital, Guangzhou, Guangdong